CLINICAL TRIAL: NCT03732768
Title: A Phase 1 Study to Evaluate the Dose, Safety and Tolerability of an Intraperitoneal α-emitting Radionuclide Therapy (Radspherin®) in Patients With Platinum Sensitive Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma With Peritoneal Carcinomatosis Following CRS
Brief Title: Study of Radspherin® in Recurrent Ovarian Cancer Subjects With Peritoneal Carcinomatosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oncoinvent AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RAD-18-001; 2018-002802-29 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Peritoneal Carcinomatosis; Ovarian Cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study followed by an expansion cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radspherin (Experimental)
  Interventions: Drug: Radspherin

INTERVENTIONS:
Drug: Radspherin — Radspherin® suspension consists of bio-degradable calcium carbonate micro particles with the α-emitting radionuclide 224Ra in suspension. 224Ra has a physical half-life of 3.6 days. The Sponsor will provide Radspherin® in single dose glass vial and the dose for each subject will be prepared at the site.

SUMMARY:
RAD-18-001 is a First-In-Man, Dose Escalation study conducted at 2 sites. The dose escalation will be performed based on a 3 + 3 design. Increasing dose levels starting at 1 MBq will be followed by 2, 4 and 7 MBq. If the highest dose level of 7 MBq is reached without Dose Limiting Toxicicities (which will stop the dose escalation), this will be the recommended dose for further exploration. Each subject will be followed until disease progression (in the abdominal cavity), or for 24 months after the administration of Radspherin® (whichever comes first).

In the expansion cohort the subject will receive the recommended dose. The expansion cohort will be conducted at 4 sites. Each subject will be followed until disease progression (in the abdominal cavity), or for 24 months after the administration of Radspherin® (whichever comes first).

DETAILED DESCRIPTION:
The maximum number of subjects enrolled in this study is 49.

The following number of subjects will be recruited in the different cohorts:

* Dose escalation cohorts: 3 - 24 Subjects
* Expansion cohort: Up to 25 Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the clinical study protocol
2. Age ≥ 18 years
3. Histologically confirmed epithelial ovarian, fallopian tube and primary peritoneal carcinoma
4. Platinum sensitive recurrences of ovarian carcinoma who are eligible for debulking surgery to R0.
5. AEs recovered to at least grade 1 from the effects (excluding alopecia) of any prior medical therapy for malignancy at time of first administration of Radspherin®
6. ECOG Performance Status Score of 0 - 1
7. Adequate renal function

   * Creatinine ≤ 1.8 mg/dl (159 μmol/l) and
   * calculated creatinine clearance using the Cockcroft-Gault formula ≥ 45 ml/min, or
   * measured creatinine clearance ≥ 45 ml/min
8. Adequate hepatic function

   * Serum bilirubin <1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
9. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/l
   * Platelets ≥ 100 x 10^9/l
   * Haemoglobin ≥ 9 g/dL
10. Adequate coagulation tests: INR ≤ 1.5 x ULN
11. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment
12. For females of childbearing potential who have a male partner: agreement to use two adequate methods of contraception (e.g. barrier, intrauterine device, hormonal implants, combined oral contraceptives or vasectomized partner), during the treatment period and for at least 3 months after the last dose of IMP.

Exclusion Criteria:

1. Neuroendocrine tumors, or non-epithelial ovarian cancers (e.g. germ cell tumors, Sex-cord tumors)
2. Tumors of borderline malignancy
3. Other synchronous visceral metastatic lesions, symptomatic CNS metastases. Metastatic lymph nodes are acceptable, except thoracic lymph nodes.
4. Pregnant or lactating (nursing) women
5. Active infections requiring antibiotics, and/or physician monitoring or recurrent fever >38.0 ⁰C associated with a clinical diagnosis of active infection
6. Active liver disease with positive serology for active hepatitis B, hepatitis C or known HIV
7. Administration of an investigational medicinal product within 28 days, or at least 5 times the half-life, prior to enrolment
8. Concurrent administration of any cancer therapy other than planned study treatment within 4 weeks prior to, and up to 4 weeks after the last study treatment
9. Another primary malignancy within the past 3 years (except for non-melanoma skin cancer, cervical cancer in situ or in situ stage 1 synchronous endometrial cancer)
10. Concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/IV cardiac disease
11. Any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise the safety of the subjects or interfere with the evaluation of the safety of the IMP
12. In the Investigator's opinion not able to comply with study procedures. Any medical or psychological condition that would preclude participation in the study or compromise the ability to give informed consent
13. Treatment with bevacizumab (Avastin®) within 5 weeks prior to CRS
14. Known hypersensitivity to any of the excipients in the study drug
15. Persons who have been placed in an institution under an official or judicial order
16. Persons who are dependent on the sponsor financially must be excluded from participation
17. Persons with active SARS-CoV-2 infection must be excluded from participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity (Ovarian Cancer)
Enrollment: 49 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities as assessed by CTCAE v5.0. | 24 months
  To investigate safety and toxicity of Radspherin®
Maximum Tolerated Dose (MTD) | 21 days
  To determine the MTD of Radspherin®, among the four suggested doses 1, 2, 4 and 7 MBq, as a single intraperitoneal (IP) injection and two repeated IP injections following cytoreductive surgery (CRS)

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven, Leuven, Belgium
- The Norwegian Radiumhospital, Oslo, Norway
- Spain (2):
  - Clínica Universidad de Navarra, Madrid
  - Clínica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Van Nieuwenhuysen E, Revheim ME, Deroose CM, Eriksson AGZ, Eyjolfsdottir B, Van Gorp T, Baert T, Aksnes AK, Myren K, Vergote I, Bruland OS. First experience with intraperitoneal 224Ra-labeled microparticles after cytoreductive surgery in patients with peritoneal recurrence of platinum-sensitive epithelial ovarian cancer. Gynecol Oncol. 2026 Jan;204:158-164. doi: 10.1016/j.ygyno.2025.11.018. Epub 2025 Dec 4. PMID 41349345